CLINICAL TRIAL: NCT05013424
Title: A Phase 2a Multicenter Open-label Study to Evaluate the Safety and Efficacy of OnabotulinumtoxinA X in Subjects With Glabellar Lines
Brief Title: A Study of OnabotulinumtoxinA X Injection in Adult Participants With Glabellar Lines
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M21-324
Record Dates: First submitted 2021-08-13; First posted 2021-08-19 (Actual); Results first posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Glabellar Lines
Keywords: Glabellar Lines; OnabotulinumtoxinA X; BOTOX
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Formulation A: OnabotulinumtoxinA (Experimental): Participants will receive one dose of OnabotA X administered as 5 injections to the corrugator and procerus muscles on Day 1.
  Interventions: Drug: Formulation A: OnabotulinumtoxinA
- Formulation B: OnabotulinumtoxinA (Experimental): Participants will receive one dose of OnabotA X administered as 5 injections to the corrugator and procerus muscles on Day 1.
  Interventions: Drug: Formulation B: OnabotulinumtoxinA
- Formulation C: OnabotulinumtoxinA (Experimental): Participants will receive one dose of OnabotA X administered as 5 injections to the corrugator and procerus muscles on Day 1.
  Interventions: Drug: Formulation C: OnabotulinumtoxinA

INTERVENTIONS:
Drug: Formulation A: OnabotulinumtoxinA — Intramuscular Injection
  Other Names: BOTOX; OnabotulinumtoxinA
  Arms: Formulation A: OnabotulinumtoxinA
Drug: Formulation B: OnabotulinumtoxinA — Intramuscular Injection
  Other Names: BOTOX
  Arms: Formulation B: OnabotulinumtoxinA
Drug: Formulation C: OnabotulinumtoxinA — Intramuscular Injection
  Other Names: BOTOX
  Arms: Formulation C: OnabotulinumtoxinA

SUMMARY:
Hyperfunctional facial lines that develop from repeated facial expression, such as glabellar lines (GL), are typically treated by selectively weakening specific muscles with small quantities of botulinum toxin. BOTOX (onabotulinumtoxinA) was first approved for aesthetic treatment of glabellar lines in 2001 and is one of the most common nonsurgical procedures in aesthetic medicine. This is a proof-of-concept study to evaluate how safe this new OnabotA X formulation is in treating adult participants with GL .

OnabotA X is an onabotulinumtoxinA investigational product being developed for the treatment of moderate to severe glabellar lines (GL). This is a 180-day, open-label study to assess the safety of a single dose of 3 different formulations of OnabotA X (A, B & C; each with varying amounts of the standard excipients in the formulation) in adult subjects with moderate to severe GL. Around 90 participants will be enrolled in the study in approximately 5 sites in the United States.

Participants will receive one dose of OnabotA X administered as 5 injections on Day 1.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular weekly visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Participant has sufficient visual acuity without the use of eyeglasses (contact lens use is acceptable) to accurately assess their facial lines.
* Participant has severe GL at maximum frown as assessed by both the investigator and participant using the Facial Wrinkle Scale - Glabellar Lines (FWS-GL) at Baseline.

Exclusion Criteria:

* History of known immunization to any botulinum toxin serotype.
* History of known hypersensitivity to any botulinum toxin serotype, or any other constituents of the study drug or its excipients, and/or other products in the same class.
* Presence or history of any medical condition that may place the participant at increased risk following exposure to OnabotA X or interfere with the study evaluation, including:

  * Diagnosed myasthenia gravis, Lambert-Eaton syndrome, amyotrophic lateral sclerosis, or any other significant disease that might interfere with neuromuscular function
  * History of facial nerve palsy
  * Infection or dermatological condition at the site of study drug injection
  * Marked facial asymmetry, dermatochalasis, deep dermal scarring, excessively thick sebaceous skin, excessively photodamaged skin, or the inability to substantially lessen facial lines even by physically spreading them apart
  * Any eyebrow or eyelid ptosis at baseline or Day 1 as determined by the investigator

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-07-07 (Actual); Study Completion 2022-07-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ALLERGAN INC., Study Director — Allergan
Locations (5):
- United States (5):
  - Advanced Research Associates - Glendale /ID# 227368, Glendale, Arizona
  - Skin Research Institute LLC /ID# 227366, Coral Gables, Florida
  - Etre Cosmetic Dermatology and Laser Center /ID# 227365, New Orleans, Louisiana
  - The Center for Dermatology Cosmetics & Laser Surgery /ID# 227369, Mount Kisco, New York
  - Austin Institute for Clinical Research /ID# 227367, Pflugerville, Texas

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Formulation A: OnabotulinumtoxinA | Formulation B: OnabotulinumtoxinA | Formulation C: OnabotulinumtoxinA
Started | 29 | 32 | 31
Completed | 28 | 30 | 30
Not Completed | 1 | 2 | 1
Not completed — Lost to Follow-up | 1 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized subjects who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Formulation A: OnabotulinumtoxinA | Formulation B: OnabotulinumtoxinA | Formulation C: OnabotulinumtoxinA | Total
Number analyzed (Participants) | 29 | 31 | 31 | 91
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.2 (11.47) | 45.7 (9.97) | 49.4 (9.96) | 49.0 (10.69)
Age, Customized [Number; unit: participants]
  18-25 years | 1 | 2 | 0 | 3
  26-40 years | 3 | 6 | 7 | 16
  41-55 years | 12 | 18 | 15 | 45
  56-64 years | 10 | 3 | 8 | 21
  >=65 years | 3 | 2 | 1 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 31 | 31 | 91
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 8 | 6 | 19
  Not Hispanic or Latino | 24 | 23 | 25 | 72
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Participants who reported multiple races are only included in 'Multiple' category.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0
    Asian | 0 | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Black or African American | 2 | 0 | 2 | 4
    White | 27 | 31 | 28 | 86
    More than one race | 0 | 0 | 1 | 1
    Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a casual relationship with this treatment. The investigator assesses the relationship of each event to the use of the study. A serious adverse event (SAE) is an event that results in death, is life threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event, that based on medical judgment, may jeopardize the participant and may require medical or surgical intervention to prevent any of the outcomes listed above. Treatment-emergent adverse events/ treatment emergent serious adverse events (TEAEs/TESAEs) are defined as any event that began or worsened in severity on or after the first dose of the study drug.
Time Frame: Day 1 to Day 180
Population: All participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Formulation A: OnabotulinumtoxinA | Formulation B: OnabotulinumtoxinA | Formulation C: OnabotulinumtoxinA
Number analyzed (Participants) | 29 | 31 | 31
Participants
  Treatment-Emergent Adverse Events (TEAE) | 7 | 15 | 9
  TEAE Related to Study Treatment | 2 | 5 | 1
  TEAE Related to Study Procedure | 0 | 4 | 1
  TEAE Related to Study Drug | 2 | 3 | 1

ADVERSE EVENTS:
Time Frame: All-cause mortality and adverse event tables include events reported from the time of informed consent to the end of the study. The median time on follow-up was 188, 184.5 and 190 days for Formulation A: OnabotulinumtoxinA, Formulation B: OnabotulinumtoxinA and Formulation C: OnabotulinumtoxinA, respectively.
Groups:
- Formulation B: OnabotulinumtoxinA; Formulation C: OnabotulinumtoxinA: Participants will receive one dose of OnabotA X administered as 5 injections to the corrugator and procerus muscles on Day 1.
  Formulation A: OnabotulinumtoxinA: Intramuscular Injection
Arm/Group | Formulation A: OnabotulinumtoxinA | Formulation B: OnabotulinumtoxinA | Formulation C: OnabotulinumtoxinA
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/32 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/29 | 1/32 | 0/31
Other Adverse Events (participants affected / at risk) | 4/29 | 9/32 | 7/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Formulation A: OnabotulinumtoxinA (N=29) | Formulation B: OnabotulinumtoxinA (N=32) | Formulation C: OnabotulinumtoxinA (N=31)
HYPERTENSIVE URGENCY (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Formulation A: OnabotulinumtoxinA (N=29) | Formulation B: OnabotulinumtoxinA (N=32) | Formulation C: OnabotulinumtoxinA (N=31)
INJECTION SITE PRURITUS (General disorders) | 2 (2) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 6 (6) | 6 (6)
URINARY TRACT INFECTION (Infections and infestations) | 2 (3) | 3 (3) | 3 (4)
HEADACHE (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2021-09-07): https://cdn.clinicaltrials.gov/large-docs/24/NCT05013424/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-02): https://cdn.clinicaltrials.gov/large-docs/24/NCT05013424/SAP_001.pdf